CLINICAL TRIAL: NCT04984148
Title: Construction of CT Radiomics Model to Assess PD-L1 Status and Predict the Efficacy of Chemoradiotherapy Combined With Immunotherapy in Unresectable Locally Advanced Non-small Cell Lung Cancer
Brief Title: Construction of CT Radiomics Model for Predicting the Efficacy of Immunotherapy in Patients With Stage III NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Shenzhen University (Other)
Responsible Party: Principal Investigator, YI PAN, Head of the Department of Radiation Oncology, Guangdong Provincial People's Hospital
Other Study IDs: GDREC2019152H
Record Dates: First submitted 2021-07-25; First posted 2021-07-30 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Stage III Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; radiomics; immunotherapy; chemoradiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trial cohort：Chemoradiotherapy followed by immunotherapy: Contrast-enhanced thoracic CT: before, during and after radiotherapy
  Radiomics
  PD-L1 testing (Histological analysis of biopsy)
  Molecular Markers (Histological analysis of biopsy)
  Interventions: Diagnostic Test: CT

INTERVENTIONS:
Diagnostic Test: CT — Contrast-enhanced thoracic computed tomography
  Other Names: Radiomics

SUMMARY:
Consolidation immunotherapy of immune checkpoint inhibitor (ICI) following chemoradiotherapy (CRT) is the current standard of care for patients with unresectable locally advanced non-small cell lung cancer (NSCLC) as it improves both progression-free survival and overall survival. However, a substantial proportion of patients still experience disease recurrence despite consolidation ICI. It is important for personalized treatment to predict the efficacy of consolidation ICI. PD-L1 expression is used as a predictive biomarker for ICI response and efficacy in advanced NSCLC, but its role in patients with stage III disease is unclear. One important reason is PD-L1 testing performed on pre-CRT tissue may not reflect changes in PD-L1 expression after CRT. CT-based radiomics approaches have been successfully applied to generate imaging biomarkers as decision support tools for clinical practice. The hypothesis of this study is that CT radiomics model can assess PD-L1 status after CRT and predict the efficacy of CRT combined with ICI in unresectable locally advanced NSCLC.

DETAILED DESCRIPTION:
This is an observational longitudinal prospective study.

CT scan is performed before radiotherapy, during radiotherapy and at the end of radiotherapy in patients with unresectable locally advanced NSCLC who undergo CRT. Radiomic features were extracted from CT images and baseline PD-L1 expression is assessed. CT-based radiomics models is developed to assess PD-L1 expression and predict the efficacy of ICI.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proven non-small cell lung cancer
* Unresectable stage III according to American Joint Committee of Cancer stage (the eighth edition)
* 18 years or older

Exclusion Criteria:

* Previous thoracic radiotherapy
* Palliative treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with stage III NSCLC undergo radical intervention.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
The association of CT radiomics features with PD-L1 expression of the tumor | 12 weeks
  To construct a radiomics model for predicting PD-L1 expression after chemoradiotherapy

SECONDARY OUTCOMES:
Association between CT radiomics model and progression-free survival of chemoradiotherapy followed by ICI | From date of inclusion to the trial until the date of first documented iRECIST progression or date of death from any cause, assessed up to 5 years
  To construct CT radiomics model for evaluating progression-free survival in patients undergo chemoradiotherapy followed by ICI
Association between CT radiomics model and overall survival of chemoradiotherapy followed by ICI | From date of inclusion to the trial until the date of death from any cause, assessed up to 5 years
  to assess the association between CT radiomics features and overall survival
Association between CT radiomics model and ICI related pneumonitis | 5 years
  To develop CT radiomics signatures for predicting ICI related pneumonitis

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China